CLINICAL TRIAL: NCT05694624
Title: Investigations Into the Mechanisms for Bioenergetic Failure in Sepsis-associated Acute Kidney Injury
Brief Title: Investigations Into Sepsis-associated Acute Kidney Injury
Status: Recruiting | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: Record ID 3055
Record Dates: First submitted 2022-12-05; First posted 2023-01-23 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — p-Aminohippuric Acid; Iohexol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis patients: Patients admitted to the intensive care unit with sepsis diagnosed or suspected
  Interventions: Drug: Para Aminohippurate
- Surgical patients: Previously healthy patients who are operated for colon cancer with laparoscopic technique.
  Interventions: Drug: Para Aminohippurate

INTERVENTIONS:
Drug: Para Aminohippurate — Measurements of renal plasma flow and glomerular filtration rate
  Other Names: iohexol

SUMMARY:
In this study the investigators would like to study systemic and regional disturbances in patients with sepsis-associated acute kidney injury and in healthy controls undergoing laparoscopic abdominal surgery. Specifically study metabolic, hemodynamic and oxygen transport variables.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) in patients with sepsis has a very poor prognosis with up to 60% mortality. The pathobiology remains to be fully understood. Creatine and phosphocreatine, products of arginine metabolism through L-arginine:glycine amidinotransferase (AGAT) and its sister enzyme guanidinoacetate N-methyl-transferase (GAMT), provide an energy-buffering system that is essential for intracellular adenosine triphosphate (ATP) supply. We hypothesized that sepsis associated AKI may be caused by failure of this energy-buffering system. In series of pilot studies, we explored metabolic and bioenergetic patterns in patients and animals with high risk of developing AKI. These data suggest that sepsis associated AKI may be caused by failure of this alternative renal energy source. In the current application we propose a clinical investigation of renal metabolism and renal bioenergetics in patients with high and low risk of developing sepsis associated AKI. The primary objective is to directly investigate renal AGAT activity through the arginyl metabolites homoarginine, guanidino acetate, and creatine. Secondary objectives are to study renal and systemic hemodynamics, renal oxygenation, glomerular filtration rate (GFR), renal tubular function, and mitochondrial respiration.

ELIGIBILITY:
Inclusion Criteria sepsis group:

* Sepsis diagnosed or suspected
* Normal premorbid serum creatinine measured or anticipated (if data are not available)
* Normovolemia as indicated by a pulse pressure variation less than 12%

Comparator group

* Previously healthy individuals scheduled for laparoscopic colon cancer resection
* Normal creatinine levels within 3 months before admittance to hospital.

  * Patients admitted to the intensive care unit with sepsis diagnosed or suspected
  * Previously healthy patients listed for elective colon cancer surgery

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensiv care patients Surgical patients
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemodynamics | Repeated measures at 10am, 12am, 2pm, 4pm,6pm, and 8pm
  Systemic and regional hemodynamics

SECONDARY OUTCOMES:
Metabolic alterations | Repeated measures at 10am, 12am, 2pm, 4pm,6pm, and 8pm
  Renal arginine metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Lars MG Ytrebø, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No